CLINICAL TRIAL: NCT04297748
Title: A Bioimaging Study of 89Zr-M7824 PET Scans in Patients With Advanced or Metastatic NSCLC Receiving M7824 Alone or in Combination With Chemotherapy
Brief Title: Bioimaging Study of 89Zr-M7824 in NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Efficacy finding
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Merck Healthcare KGaA (Unknown); Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2018-001
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: PD-L1; TGF-beta; 89Zr-PET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Camurati-Engelmann Syndrome | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Intervention Model Description: The study will enroll into two sequential cohorts A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients (pts) will receive an initial trace (100 mg, IV) dose of zirconium-89 (1.8-2.5 mCi) labelled M7824 (89Zr-M7824) on day 1, sequential PET imaging over 1 week will be performed to determine the biodistribution 89Zr-M7824 into the tumour and normal tissues. All patients who remain on study after Day 14 will have a 1200 mg dose of M7824 q2w beginning on Cycle 1 Day 15. Pts will then receive a 2nd infusion of 100 mg of 89Zr-M7824 with cold M7824 making a total dose of 1200mg on Day 29. All patients will then receive a dose of cold 1200mg M7824 on Cycle 1 Day 43. Patients will continue to receive a therapeutic dose of 1200 mg q2w of M7824 until disease progression or unacceptable toxicity. Patients who do not achieve a CR after 3 doses of M7824 in Cycle 1, may then commence treatment with concurrent chemotherapy with carboplatin and pemetrexed at conventional doses.
  Interventions: Combination Product: 89Zirconium-M7824; Drug: M7824
- Cohort B (Experimental): Cohort A will determine whether or not high PD-L1 positive disease is required at study entry to Cohort B. All other assessments within cohort A will be undertaken.
  Interventions: Combination Product: 89Zirconium-M7824; Drug: M7824

INTERVENTIONS:
Combination Product: 89Zirconium-M7824 — PET imaging agent
Drug: M7824 — Bifunctional fusion protein intended to block PD-L1 and neutralize TGFbeta simultaneously.
  Other Names: bintrafusp alfa

SUMMARY:
This is a bioimaging study of 89Zr-M7824 PET scans in patients with advanced or metastatic non-small cell lung cancer who will be receiving M7824 alone or with standard of care chemotherapy. M7824 is a bifunctional fusion protein that combines an anti-PD-L1 antibody and the extracellular domain of TGFβ receptor II (TGFβRII) as a TGFβ neutralizing 'trap', into a single molecule.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors have shown improved treatment outcome in patients with NSCLC; however, there is room to further improve benefits. A novel agent such as M7824, a fusion protein which targets the tumor microenvironment where it blocks both the cell intrinsic PD-L1/PD-1 interaction and the immunosuppressive TGFβ, is hypothesized to be more effective than agents that target only a single pathway.

This study aims to investigate functional imaging with 89Zr-M7824 to characterize the biodistribution of M7824 to support its clinical development. In Part A, we will evaluate the biodistribution of zirconium-89 (89Zr) labelled M7824 in a small cohort of lung cancer patients unselected for PD-L1 status (n=3). In particular, we will examine the ability of 89Zr-M7824 to detect and quantitate intra-tumoural PD-L1 expression and correlate this with PD-L1 assessment in archival tissue. Based on this, Part B will gather additional data about the biodistribution of 89Zr-M7824 in an additional 9 patients. The requirement for patients in Part B to have high levels of PD-L1 positive cells in tumours based on a fresh biopsy or archival tissue at study entry will be informed by the data generated in Part A. Safety will be formally assessed also as a secondary endpoint at the end of Part A of the study and addressed if necessary. After completion of 2 imaging cycles, patients who do not show complete response to M7824 monotherapy after 3 therapeutic doses of M7824 may be transitioned to M7824/chemotherapy combination

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) with histologically proven advanced NSCLC
* PD-L1 positive staining in > 1% of tumour cells in archival or fresh tissue (may be modified for Cohort B to require PDL1-high status and/or PD-L1 status to be tested on fresh tissue obtained a study entry, based on evaluation of data from Cohort A)
* Measurable disease by RECIST 1.1
* ECOG 0-1
* Expected survival more than 3 months
* Adequate organ function. Out of range values that are not clinically significant will be permitted, except for the following laboratory parameters, which must be within the ranges specified:

Hemoglobin ≥ 9 g/dL Neutrophils ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L INR ≤ 1.4 Serum creatinine ≤1.3 x ULN Estimated creatinine clearance ≥ 30 ml/min according to the Cockcroft Gault formula or local normal range Serum AST and ALT ≤2.5 x ULN Serum bilirubin ≤ 1.5 x ULN Available archived formalin-fixed paraffin embedded or frozen tumour tissue; or consents to tumour biopsy at enrolment (the latter is strongly preferred) Presence of a suitable reference tumour lesion for PET imaging i.e. measuring > 1.5cm and not located in the mediastinum

Exclusion Criteria:

* Prior systemic immunotherapy for advanced NSCLC
* Patients who are unsuitable for chemotherapy in the investigator's judgement
* The participant's tumour harbors an EGFR sensitizing (activating) mutation, ALK translocation, ROS1 rearrangement, or BRAF V600E mutation
* Use of anti-cancer therapy including surgery, chemotherapy, immunotherapy, radiotherapy to a non-thoracic site or any investigational therapy within 28 days prior to Study Day 1
* Has received thoracic radiotherapy > 30 Gy within 6 months of the dose of study drug
* Previous malignant disease (other than NSCLC) within the last 3 years. Participants with a history of cervical carcinoma in situ, superficial or non-invasive bladder cancer, or basal cell or squamous cell carcinoma in situ previously treated with curative intent are NOT excluded. Participants with other localized malignancies treated with curative intent need to be discussed with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 89Zr-M7824 in NSCLC patients | Cycle 1 - 7 weeks
  The biodistribution of 89Zr-M7824 will be evaluated by qualitative assessment of organ uptake and clearance from PET imaging following infusion of 89Zr-M7824. Patterns of expected normal tissue uptake due to blood pool activity, and PD-L1 expression, as well as catabolism of 89Zr-M7824, will be assessed.

SECONDARY OUTCOMES:
Number of participants with 89Zr-M7824 treatment-related adverse events as assessed using CTCAE v5.0. | 0-12 months
  Adverse responses of any grade following commencement of treatment will be recorded and quantified.
Number of participants with M7824 or M7824 combined with chemotherapy treatment-related adverse events as assessed using CTCAE v5.0. | 0-36 months
  Adverse responses of any grade following commencement of treatment will be recorded and quantified.

OTHER OUTCOMES:
Clinical outcomes assessed via response evaluation criteria in solid tumors (RECIST) V1.1 | 0-36 months
  Describe response rates to M7824 monotherapy or M7824 combined with conventional chemotherapy, defined as number of patient achieving a complete disease response, partial disease response or stable disease response determined by medical imaging of tumours.
Correlation of clinical outcome of monotherapy with M7824 (assessed via RECIST) with tumour uptake of 89Zr-M7824 as quantified by PET imaging. | 0-12 months
  To determine association of response to M7824 monotherapy with tumour uptake of 89Zr-M7824.
Quantification of PD-L1 expression IHC and tumour uptake in a given lesion as measured by 89Zr-M7824 biodistribution. | 0-12 months
  To determine the association between PD-L1 expression determined by IHC and tumour uptake in a given lesion as measured by 89Zr-M7824 biodistribution.

CONTACTS AND LOCATIONS:
Overall Officials: Hui K Gan, MBBS, Principal Investigator — Austin Health; Andrew M Scott, MBBS, Principal Investigator — Austin Health
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No